CLINICAL TRIAL: NCT04762277
Title: Randomized, Double-blind, Placebo-controlled, Study of Spesolimab in Patients With Moderate to Severe Hidradenitis Suppurativa
Brief Title: A Study to Test Whether Spesolimab Helps People With a Skin Disease Called Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1368-0052; 2020-003672-40 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spesolimab (Experimental)
  Interventions: Drug: Spesolimab - solution for infusion; Drug: Spesolimab- solution for injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching spesolimab - solution for infusion; Drug: Placebo matching to spesolimab- solution for injection

INTERVENTIONS:
Drug: Spesolimab - solution for infusion — Solution for infusion
  Arms: Spesolimab
Drug: Placebo matching spesolimab - solution for infusion — Solution for infusion
  Arms: Placebo
Drug: Spesolimab- solution for injection — Solution for injection
  Arms: Spesolimab
Drug: Placebo matching to spesolimab- solution for injection — Solution for injection
  Arms: Placebo

SUMMARY:
This study is open to adults with a chronic inflammatory skin disease called hidradenitis suppurativa. The purpose of this study is to find out whether a medicine called spesolimab helps people with moderate to severe hidradenitis suppurativa.

Participants are put into 2 groups by chance. One group takes spesolimab. The other group takes placebo. Every participant has twice the chance of being in the spesolimab group than in the placebo group. Participants get spesolimab or placebo as an infusion into a vein every week for the first 3 weeks. Afterwards, they get spesolimab or placebo as injections under the skin every 2 weeks. Placebo infusions and injections look like spesolimab infusions and injections but do not contain any medicine.

Participants are treated in the study for about 3 months. During this time, they visit the study site about 9 times. After completing this part of the study, participants are offered to join another clinical study in which all participants get spesolimab. Participants who cannot join the other study, stay in this study for about 4 more months. During this time, participants do not take spesolimab nor placebo but they visit the study site 2 times to have their health checked.

At study visits, doctors thoroughly check the skin of participants to count lumps (nodules) and boils (abscesses). The results between the spesolimab group and the placebo group are compared after 3 months of treatment. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patients, 18 years of age or older
* Signed and dated written informed consent in accordance with International Council on Harmonisation (ICH) Good Clinical Practice (GCP) and local legislation prior to the start of any screening procedures
* Moderate to severe Hidradenitis suppurativa (HS), based on International Hidradenitis Suppurativa Severity Score System (IHS4) criteria, for at least 1 year prior to the baseline visit, as determined by the investigator through participant interview and/or review of the medical history. (If IHS4 scoring is not available, equivalent scoring based on scoring systems as HS-PGA or Hurley are acceptable based on documented investigator assessment)
* HS lesions in at least 2 distinct anatomic area (right/left axillary, inguinal, inframammary, perineal)
* Biologic naive or TNF inhibitor (TNFi)-failure for HS
* Inadequate response to an adequate course of appropriate oral antibiotics for treatment of HS in the last 1 year, as per investigator discretion. This is not applicable for TNFi-failure patients
* Total abscess and inflammatory nodule (AN) count of greater than or equal to 5
* Total draining fistula count of less than or equal to 20 Further inclusion criteria apply

Exclusion Criteria:

* Presence of active skin lesions other than HS that interfere with the assessment of HS
* Use of restricted medications as below:

  * Topical corticosteroids over HS lesions within 1 week of Visit 2
  * Systemic antibiotics within 4 weeks of visit 2
  * Systemic non-biologic immunomodulatory and/or immunosuppressive agents use for HS within 4 weeks (or 5 half lives, whichever is longer) of visit 2
  * Biologic agents use within 12 weeks or 5 half-lives, whichever is longer, prior to visit 2
  * Opioid analgesics within 2 weeks of visit 2
  * Live virus vaccine within 6 weeks of visit 2
* Prior exposure to any immunosuppressive biologic other than TNFi for HS
* Prior exposure to Interleukin 36 Receptor (IL-36R) inhibitors including spesolimab
* Treatment with any investigational device or investigational drug of chemical or biologic nature within a minimum of 30 days or 5 half-lives of the drug, whichever is longer, prior to visit 2
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial. Women who stop nursing before the study drug administration do not need to be excluded from participating
* History of allergy/hypersensitivity to the systemically administered trial medication agent or its excipients
* Patient with a transplanted organ (with exception of a corneal transplant > 12 weeks prior to screening) or who have ever received stem cell therapy (e.g., Remestemcel-L) Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (5):
  - Dermatology Research Associates, Los Angeles, California
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Australia (2):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Royal Melbourne Hospital, Parkville, Victoria
- ULB Hopital Erasme, Brussels, Belgium
- Dr. S. K. Siddha Medicine Professional Corporation, Newmarket, Ontario, Canada
- University Hospital Ostrava, Ostrava, Czechia
- France (3):
  - CLI Reims Bezannes, Bezannes
  - HOP Edouard Herriot, Lyon
  - HOP Larrey, Toulouse
- Germany (3):
  - Katholisches Klinikum Bochum gGmbH, Bochum
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Frankfurt, Frankfurt am Main
- Italy (2):
  - Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliera Universitaria Pisana, Pisa
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Nordlandssykehuset HF, Bodø, Bodø
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
- Poland (2):
  - Non-Public Health Care Facility LABDERM, Ossy
  - Cityclinic Medical and Psychological Clinic Matusiak Partnership, Wroclaw
- Hospital Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Lebwohl MG, Thoma C, Haeufel T. Spesolimab use in generalised pustular psoriasis flares - Authors' reply. Lancet. 2024 Aug 31;404(10455):847-848. doi: 10.1016/S0140-6736(24)01557-5. No abstract available. PMID 39216969
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an international, phase IIa multi-center, double-blind, placebo-controlled trial assessing the efficacy and safety of spesolimab in patients with moderate to severe Hidradenitis suppurativa (HS).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Patients received placebo administered intravenously (i.v.) at Weeks 0, 1, and 2, and subcutaneously injection at Weeks 4, 6, 8, and 10.
- Spesolimab: Patients received 1200 mg of spesolimab administered intravenously (i.v.) at Weeks 0, 1, and 2, and subcutaneously injection at Weeks 4, 6, 8, and 10.
Period: Overall Study
Arm/Group | Placebo | Spesolimab
Started | 17 | 35
Completed (Completed treatment) | 16 | 32
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Spesolimab | Total
Number analyzed (Participants) | 17 | 35 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (11.0) | 35.7 (11.3) | 35.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 31
  Male | 7 | 14 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 29 | 44
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 12 | 23 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Total number of abscesses and inflammatory nodules [Mean (Standard Deviation); unit: abscesses and inflammatory nodules] — Total number of abscesses and inflammatory nodules at baseline.
  abscesses and inflammatory nodules | 18.9 (15.7) | 11.6 (9.3) | 14.0 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Abscess and Inflammatory Nodule Count at Week 12
Description: Percent change from baseline in total abscess and inflammatory nodule count at Week 12= [(Total Abscess at Week 12 + Total Inflammatory Nodule at Week 12) - (Total Abscess at baseline + Total Inflammatory Nodule at baseline)] *100/ (Total Abscess at baseline + Total Inflammatory Nodule at baseline).
  Percent change from baseline in total abscess and inflammatory nodule count at Week 12 was modelled using mixed effects model for repeated measures (MMRM) accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, the effect of stratum (stratification according to tumor necrosis factor inhibitor (TNFi)-naive population vs. TNFi-failure population) and the fixed continuous effects of baseline at each visit (Weeks 1, 2, 4, 6, 8, 10, and 12). The Least Squares Mean (Standard Error) at Week 12 is reported.
Time Frame: MMRM included measurements from baseline (Week 0) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration. MMRM estimates of percent change from baseline to Week 12 is reported.
Population: Safety Analysis Set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug. Data up to use of rescue therapy were included for analysis, and data post the use were censored. Only patients with non-missing endpoint data were included.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 14 | 30
percent change | -34.7 (11.1) | -38.8 (7.5)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; MMRM accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, the effect of stratum (stratification according to TNFi-naive population vs. TNFi-failure population) and the fixed continuous effects of baseline at each visit. The unstructured covariance structure was used to model the within patient measurements. To estimate denominator degrees of freedom the Kenward-Roger approximation was used; Test type: Other; Mean Difference (Net) = -4.1, 95% CI 2-sided [-31.7 to 23.4] — Difference of Least Squares Means was calculated as: Spesolimab-Placebo

2. Secondary Outcome: Percent Change From Baseline in Draining Fistula Count at Week 12
Description: Percent change from baseline in draining fistula at Week 12 was calculated as: [(total draining fistula at Week 12) - (total draining fistula at baseline)] * 100 %/ (total draining fistula at baseline).
  Percent change from baseline in draining fistula count at Week 12 was modelled using mixed effects model for repeated measures (MMRM) accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, the effect of stratum (stratification according to tumor necrosis factor inhibitor (TNFi)-naive population vs. TNFi-failure population) and the fixed continuous effects of baseline at each visit (Weeks 1, 2, 4, 6, 8, 10, and 12). The Least Squares Mean (Standard Error) at Week 12 is reported.
Time Frame: MMRM included measurements from baseline (Week 0) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration. MMRM estimates of percent change in draining fistula from baseline to Week 12 is reported.
Population: Safety Analysis Set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug. Data up to use of rescue therapy were included for analysis, and data post the use were censored. Only patients with baseline draining fistulas >=1 and non-missing endpoint data were included.
Measure: Least Squares Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 13 | 24
percent change | 56.6 (23.0) | -40.1 (16.8)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Net) = -96.6, 95% CI 2-sided [-154.5 to -38.8] — Difference of Least Squares Means was calculated as: Spesolimab-Placebo

3. Secondary Outcome: Achievement of Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12
Description: HiSCR is defined as at least a 50% reduction in the total abscess and inflammatory nodule (AN) count with no increase in abscess count and no increase in draining fistula count relative to baseline.
  Proportion of patients with achievement of Hidradenitis Suppurativa Clinical Response (HiSCR) at Week 12 is reported. Proportion of patients with achievement of HiSCR at Week 12 was calculated as: number of patients with achievement of HiSCR at Week 12/number of patients analyzed. Proportions were rounded up to three decimal places.
Time Frame: At baseline (Week 0) and at Week 12.
Population: Safety Analysis Set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug. Any binary data collected after use of any rescue therapy was censored and then imputed using the no response imputation (NRI) method as described in the statistical analysis plan.
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 17 | 35
proportion of patients | 0.176 | 0.314
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; The difference in the proportion of patients with a response between Spesolimab and placebo was analysed using a logistic regression model. The model included treatment and stratification factor (tumor necrosis factor inhibitor (TNFi)-naive population versus TNFi-failure population) as two categorical variables; Test type: Other; Risk Difference (RD) = 0.138, 95% CI 2-sided [-0.129 to 0.339] — Risk difference was calculated as: Spesolimab - Placebo. 95% Confidence Interval (CI) for treatment difference is calculated by Chan and Zhang method

4. Secondary Outcome: Absolute Change From Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) Value at Week 12
Description: The IHS4 assesses the hidradenitis suppurativa (HS) severity and the resulting IHS4 score is arrived at by= number of nodules * 1 + number of abscesses * 2 + number of draining fistula * 4.
  A total score of 3 or less signifies mild, 4-10 signifies moderate and 11 or higher signifies severe disease.
  Absolute change from baseline in IHS4 value at Week 12 was modelled using mixed effects model for repeated measures (MMRM) accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, the effect of stratum (stratification according to tumor necrosis factor inhibitor (TNFi)-naive population vs. TNFi-failure population) and the fixed continuous effects of baseline at each visit (Weeks 1, 2, 4, 6, 8, 10, and 12). The Least Squares Mean (Standard Error) at Week 12 is reported.
Time Frame: MMRM included measurements at baseline (Week 0) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration. MMRM estimates of absolute change in IHS4 from baseline to Week 12 is reported.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 14 | 30
units on a scale | 4.9 (4.7) | -9.0 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Net) = -13.9, 95% CI 2-sided [-25.6 to -2.3] — Difference of Least Squares Means was calculated as: Spesolimab-Placebo

5. Secondary Outcome: Absolute Change From Baseline in Hidradenitis Suppurativa Area and Severity Index (HASI) Score at Week 12
Description: HASI includes four domains to assess the severity of HS disease activity, which are erythema, induration, open ulcer and draining fistula and scored on a Likert scale 0 (none) to 3 (severe/extensive) for each predetermined body region.
  For body surface area (BSA) assessment, the number of palms (one palm indicates 1% of the patient's BSA) involved for each body region (head, right axilla, left axilla, anterior chest, back, anterior bathing trunk, posterior bathing trunk, other) is assessed and converted to a percentage of that region. An area score was assigned to each region using the approach (0 = none, 1 = 1-9%, 2 = 10-29%, 3 = 30-49%, 4 = 50-69%, 5 = 70-89%, 6 = 90- 100%). Scores for the four domains of HS are summed and adjusted for the area affected, and the score of each area are summed to calculate the total HASI score, which ranges from 0 (no disease) to 72 (severe disease).
  The Least Squares Mean (Standard Error (SE)) derive from MMRM.
Time Frame: MMRM included measurements at baseline (Week 0) and at Weeks 1, 2, 4, 6, 8, 10, and 12 after first drug administration. MMRM estimates of absolute change from baseline in HASI score at Week 12 is reported in the table below.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 14 | 30
units on a scale | -3.8 (6.9) | -23.6 (4.7)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Net) = -19.8, 95% CI 2-sided [-36.9 to -2.7] — Difference of Least Squares Means was calculated as : Spesolimab- Placebo

6. Secondary Outcome: Achievement of Hidradenitis Suppurativa Physician Global Assessment (HS-PGA) Score of 0 or 1 at Week 12
Description: HS-PGA documents the physician's assessment of the patient's HS at a given timepoint. The HS-PGA score ranges from 0 to 5, where: 0=clear - no abscesses, draining fistula, inflammatory nodules or noninflammatory nodules); 1=minimal - no abscesses, draining fistula or inflammatory nodules and the presence of noninflammatory nodules); 2=mild - no abscesses or draining fistula and 1-4 inflammatory nodules, or 1 abscess or draining tunnel and no inflammatory nodules); 3=moderate - no abscesses or draining fistula and ≥5 inflammatory nodules, or 1 abscess or draining fistula and ≥1 inflammatory nodule, or 2-5 abscesses or draining fistula and <10 inflammatory nodules); 4=severe - 2-5 abscesses or draining fistula and ≥10 inflammatory nodules); 5=very severe - >5 abscesses or draining fistula). Proportion of patients with achievement of HS-PGA score of 0 or 1 at Week 12 was calculated as: number of patients with achievement of HS-PGA score of 0 or 1 at Week 12/number of patients analyzed.
Time Frame: At Week 12.
Population: as for outcome 3
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 17 | 35
proportion of patients | 0.000 | 0.057
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = 0.057, 95% CI 2-sided [-0.132 to 0.186] — Risk difference was calculated as: Spesolimab-Placebo. 95% Confidence Interval (CI) for treatment difference is calculated by Chan and Zhang method

7. Secondary Outcome: Achievement of at Least 30% Reduction From Baseline in Numerical Rating Scale (NRS30) in Patient's Global Assessment of HS Pain at Week 12
Description: The HS Pain Numerical Rating Scale (NRS) is an endpoint for the assessment of HS-related pain severity. Recall period is 24 hours and response is given by an 11-point scale ranging from 0 (no pain) to 10 (worst possible pain).
  For the analysis of pain, weekly average of daily assessment was calculated for each visit based on values prior to the visit. Missing daily values within a week were ignored if there are at least 4 reported values.
  Proportion of patients with achievement of at least 30% reduction from baseline in NRS30 in Patient's Global Assessment of HS Pain at Week 12. Proportion of patients with achievement of at least 30% reduction from baseline in NRS30 in Patient's Global Assessment of HS Pain at Week 12 was calculated as: number of patients with achievement of at least 30% reduction from baseline in NRS30 in Patient's Global Assessment of HS Pain at Week 12/number of patients analyzed. Proportions were rounded up to three decimal places.
Time Frame: At baseline (Week 0) and at Week 12.
Population: as for outcome 3
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 17 | 35
proportion of patients | 0.059 | 0.229
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = 0.170, 95% CI 2-sided [-0.067 to 0.338] — Risk Difference was calculated as: Spesolimab - Placebo. 95% Confidence Interval (CI) for treatment difference was calculated by Chan and Zhang method

8. Secondary Outcome: Occurrence of Complete Elimination of Draining Fistulas at Week 12
Description: Proportion of patients with occurrence of complete elimination of draining fistulas at Week 12 is reported. Proportion of patients with occurrence of complete elimination of draining fistulas at Week 12 was calculated as: number of patients with occurrence of complete elimination of draining fistulas at Week 12/number of patients analyzed. Proportions were rounded up to three decimal places.
Time Frame: Baseline (Week 0) and at Week 12.
Population: Safety Analysis Set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug. Any binary data collected after use of any rescue therapy was censored and then imputed using the no response imputation (NRI) method as described in the statistical analysis plan. Only patients with baseline draining fistulas >= 1 and non-missing endpoint data were included.
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 15 | 28
proportion of patients | 0.067 | 0.250
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = 0.183, 95% CI 2-sided [-0.079 to 0.375] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Occurrence of at Least One Flare at Week 12
Description: Proportion of patients with occurrence of at least one flare at Week 12. Flare was defined as at least 25 % increase in abscess and inflammatory nodule count with a minimum increase of 2 relative to baseline.
  Proportion of patients with occurrence of at least one flare at Week 12 was calculated as: number of patients with occurrence of at least one flare at Week 12/number of patients analyzed. Proportions were rounded up to three decimal places.
Time Frame: At Week 12.
Population: as for outcome 3
Measure: Number; unit: proportion of patients
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 17 | 35
proportion of patients | 0.176 | 0.086
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 3, analysis 1]; Test type: Other; Risk Difference (RD) = -0.091, 95% CI 2-sided [-0.331 to 0.089] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Absolute Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI is a patient-administered, ten-question, quality of life questionnaire that covers six domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Response categories include "not relevant" (score of 0), "not at all" (score of 0), "a little" (score of 1), "a lot" (score of 2) and "very much" (score of 3). DLQI total score is calculated by summing the scores of each question resulting in a range of 0 to 30 with higher scores indicating greater health-related quality of life impairment. Absolute change from baseline in DLQI score at Week 12 was modelled using MMRM accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, the effect of stratum (stratification according to tumor necrosis factor inhibitor (TNFi)-naive population vs. TNFi-failure population) and the fixed continuous effects of baseline at each visit (Weeks 1, 4, 8, and 12).
Time Frame: MMRM included measurements at baseline (Week 0) and at Weeks 1, 4, 8, and 12 after first drug administration. MMRM estimates of absolute change in DLQI from baseline to Week 12 is reported.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 14 | 30
units on a scale | -2.8 (1.8) | -2.8 (1.2)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Net) = -0.1, 95% CI 2-sided [-4.4 to 4.3] — Difference of Least Squares Means was calculated as: Spesolimab-Placebo

11. Secondary Outcome: Absolute Change From Baseline in Hidradenitis Suppurativa Quality of Life (HiS-QoL) Total Score at Week 12
Description: HiS-QoL is a patient-administered, 17-item instrument to measure HS-specific quality of life in clinical trials with a 7-day recall period. The 17-item HiS-QoL included four symptom items, eight activity-adaptation items and five psychosocial items. The item scores are summed to create a total ranging from 0 to 68, with higher scores indicating more severe impact on health-related quality of life.
  Absolute change from baseline in HiS-QoL total score at Week 12 was modelled using MMRM accounting for the following sources of variation: fixed, categorical effects of treatment at each visit, the effect of stratum (stratification according to tumor necrosis factor inhibitor (TNFi)-naive population vs. TNFi-failure population) and the fixed continuous effects of baseline at each visit (Weeks 1, 4, 8, and 12).
Time Frame: MMRM included measurements at baseline (Week 0) and at Weeks 1, 4, 8, and 12 after first drug administration. MMRM estimates of absolute change in HiS-QoL from baseline to Week 12 is reported.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 14 | 25
units on a scale | -4.5 (3.2) | -5.8 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Spesolimab; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mean Difference (Net) = -1.3, 95% CI 2-sided [-9.5 to 6.9] — Difference of Least Squares Means was calculated as: Spesolimab-Placebo

12. Secondary Outcome: The Occurrence of Treatment Emergent Adverse Events (TEAEs)
Description: Percentage of patients with occurrence of Treatment Emergent Adverse Events (TEAEs) is reported. Percentage of patients with occurrence of Treatment Emergent Adverse Events (TEAEs) was calculated as: number of patients with occurrence of TEAEs / number of patients analyzed. Percentages were rounded to one decimal place.
  Time Frame: From first drug administration until 16 weeks after last drug administration, up to 28 weeks for patients who did not to roll-over to the open-label extension (OLE) trial (trial number 1368-0067 (NCT04876391)).
  From first drug administration until Week 12 for patients who did roll-over to the open-label extension (OLE) trial (trial number 1368-0067 (NCT04876391)).
Time Frame: Up to 12 weeks for patients who did roll-over to the open-label extension (OLE) trial (trial number 1368-0067 (NCT04876391)) and up to 28 weeks who did not roll-over to the OLE trial. For details please see description.
Population: Safety Analysis Set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug. One patient randomised to receive placebo took spesolimab during the study, therefore was considered in spesolimab arm instead for safety reporting.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Spesolimab
Number analyzed (Participants) | 16 | 36
percentage of patients | 87.5 | 77.8

ADVERSE EVENTS:
Time Frame: From first drug administration until 16 weeks after last drug administration, up to 28 weeks for patients who did not to roll-over to the open-label extension (OLE) trial (trial number 1368-0067 (NCT04876391)). From first drug administration until Week 12 for patients who did roll-over to the open-label extension (OLE) trial (trial number 1368-0067 (NCT04876391)).
Description: Safety Analysis Set (SAF): This patient set included all patients who were randomized and received at least one dose of study drug. One patient randomised to receive placebo took spesolimab during the study, therefore was considered in spesolimab arm instead for safety reporting.
Arm/Group | Placebo | Spesolimab
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/36
Other Adverse Events (participants affected / at risk) | 14/16 | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Spesolimab (N=36)
Suicidal behaviour (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Spesolimab (N=36)
Arrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 4
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 4
Injection site erythema (General disorders) | 0 | 4
Injection site nodule (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 3
Injection site papule (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3
Pilonidal cyst (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Bacterial test positive (Investigations) | 1 | 1
Platelet count increased (Investigations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 4
Sciatica (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 1
Breast discomfort (Reproductive system and breast disorders) | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 1
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 2 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT04762277/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT04762277/SAP_001.pdf